CLINICAL TRIAL: NCT07265544
Title: Single-cell Multiomics and Spatiotemporal Omics Analyze the Mechanism of Liver Degenerative Disease
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Beijing Friendship Hospital (Other); Beijing YouAn Hospital (Other); Zhongnan Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2023-207
Record Dates: First submitted 2025-06-19; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Liver Neoplasm; HBV Infection; Non-alcoholic Fatty Liver Disease NAFLD; Liver Fibrosis
Keywords: single-cell multi-omics; HBV infection; liver degenerative changes
MeSH Terms: conditions — Liver Neoplasms; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal group: Age groups are divided into minors (<18 years old), young adults (18-50 years old), and the elderly (>65 years old).
  Interventions: Procedure: Collection of Preoperative Peripheral Blood; Procedure: Collection of Discarded Liver Tissue During Surgery
- Fatty liver group: Fatty liver groups are categorized based on the degree of hepatic steatosis into mild, moderate, and severe fatty liver groups.
  Interventions: Procedure: Collection of Preoperative Peripheral Blood; Procedure: Collection of Discarded Liver Tissue During Surgery
- Liver fibrosis group: Liver fibrosis groups are distinguished according to the stage of hepatic fibrosis into mild, moderate, and severe liver fibrosis groups.
  Interventions: Procedure: Collection of Preoperative Peripheral Blood; Procedure: Collection of Discarded Liver Tissue During Surgery
- hepatitis B virus infection: Patients with hepatitis B virus (HBV) infection
  Interventions: Procedure: Collection of Preoperative Peripheral Blood; Procedure: Collection of Discarded Liver Tissue During Surgery

INTERVENTIONS:
Procedure: Collection of Preoperative Peripheral Blood — Prior to surgery, 30 milliliters of peripheral blood will be drawn from the subject's upper limb.
Procedure: Collection of Discarded Liver Tissue During Surgery — From subjects undergoing hepatectomy or liver biopsy, discarded liver tissue will be collected during the surgical procedure.

SUMMARY:
The purpose of this observational study is to employ single-cell multi-omics and spatial omics technologies to characterize the spatial and immune structures within the livers of patients with fatty liver, hepatic hemangioma, focal nodular hyperplasia, liver fibrosis, cirrhosis, and HBV infection. The primary questions it aims to address are:

Investigate the mechanisms of liver degenerative changes during the processes of liver aging, fatty liver, HBV infection, liver fibrosis, and cirrhosis.

Characterize the molecular features and cellular networks at different stages of liver degeneration and identify new targets and mechanisms for the cure of the aforementioned diseases.

The study will collect peripheral blood and discarded liver tissue from patients with hepatic hemangioma, fatty liver, HBV infection, liver fibrosis, and cirrhosis who are undergoing hepatectomy or liver biopsy.

DETAILED DESCRIPTION:
Research Objectives The purpose of this study is to leverage the strengths of clinical departments to collect preoperative peripheral blood samples and liver tissue (from hepatectomy or liver biopsy) that meet the project requirements from patients with hepatic hemangioma, focal nodular hyperplasia, fatty liver, HBV infection, liver fibrosis, and cirrhosis. This initiative aims to establish a large-scale clinical liver disease sample repository comprising 160-240 cases. The study will encompass livers across different age groups (including minors under 18 years old, adults aged 18-50 years, and the elderly over 65 years old) and varying severities of fatty liver (mild, moderate, severe), HBV infection, and liver fibrosis (early, moderate, advanced [cirrhosis]). Utilizing single-cell multi-omics (such as single-cell transcriptomics and chromatin accessibility sequencing) and spatial omics sequencing technologies, the study will construct a human spatiotemporal liver degeneration-regeneration atlas covering states of homeostasis, aging, liver fibrosis, and fatty liver. By comparing phenotypes, functions, spatial distributions, and intercellular interactions of cell populations across different groups, the study aims to identify diagnostic and therapeutic targets for cell therapy, gene therapy, or other interventions. During the study, no random or protocol-driven treatments will be administered to participants. If clinically appropriate, the treating physician will make decisions and select treatment plans based on individual circumstances.

Data Collection Procedures Given that this is a multicenter, prospective, observational study, no additional visits or laboratory analyses beyond routine clinical practice are required. Physicians will determine treatment plans in accordance with instructions and local guidelines. Researchers will review patients' medical histories and laboratory reports to determine eligibility based on inclusion and exclusion criteria. Patients must sign the most recent informed consent form (ICF) approved by the IRB/IEC before data collection. In line with routine clinical practice, surgeons will prioritize clinical needs when obtaining surgical specimens, and then collect discarded clinical samples for experimental exploration and clinical data analysis. Each participant will be assigned a unique identification number, such as Fibrosis-1, Fibrosis-2, etc. All study documents (e.g., case report forms, clinical records) will use this identification number. In compliance with data privacy regulations, the use of unique identification numbers is permitted as long as they do not contain combinations of information that could identify participants (for example, the use of participants' initials and date of birth together is not allowed).

Sample Collection Demographic Data Recording: Record date of birth, gender, and initials. Medical History and Physical Examination: Include vital signs, height, weight, physical examination of all body systems; past and present medical history, including the presence of spider angiomas or palmar erythema, dull complexion, jaundice of skin and sclera, hepatic pain, and enlargement of liver, spleen, or lymph nodes.

Preoperative Peripheral Blood Collection: Draw 30 milliliters of peripheral blood from the subject's upper limb before surgery.

Collection of Discarded Liver Tissue During Surgery: From subjects undergoing hepatectomy or liver biopsy, collect discarded liver tissue during the surgical procedure.

Safety Monitoring, Reporting, and Medical Management Adverse Event (AE) Definition: An adverse event is any unfavorable medical occurrence in a patient or subject after the administration of a drug, whether or not considered related to the treatment. Adverse events can include any adverse signs (including abnormal laboratory findings), symptoms, or diseases temporally related to the use of the study drug, regardless of whether a causal relationship with the study drug is considered. Adverse events encompass both serious adverse events (SAEs) and non-serious adverse events.

SAE Definition: An SAE is a medical event occurring during a clinical study that requires hospitalization or prolongation of hospital stay, results in disability, affects the ability to work, is life-threatening or fatal, or causes congenital anomalies. These medical events include:

Events leading to death; Life-threatening events (defined as events where the subject is at immediate risk of death at the time of the event); Events requiring hospitalization or prolongation of hospital stay; Events that may result in permanent or significant disability/functional impairment/loss of ability to work; Congenital abnormalities or birth defects; Other important medical events (defined as events that pose a hazard to the subject or require intervention to prevent any of the above situations).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent form;
2. No restrictions on age and gender;
3. Patients diagnosed with hepatic hemangioma or focal nodular hyperplasia of the liver in accordance with the "Guidelines for the Diagnosis and Treatment of Focal Liver Lesions (2014 Edition)" and the "Guidelines for the Diagnosis and Treatment of Hemangiomas and Vascular Malformations (2019 Edition)";
4. Patients with hepatic hemangioma, focal nodular hyperplasia of the liver, fatty liver, HBV infection, liver fibrosis, and cirrhosis who clinically require liver surgery or liver biopsy.

Exclusion Criteria:

1. Individuals with concurrent infections such as HIV will be excluded.
2. Patients with coagulation system disorders, such as hemophilia or idiopathic thrombocytopenic purpura, will not be included.
3. Those with severe underlying diseases that affect the body's immune status will be excluded.
4. Individuals whom the investigator deems unsuitable for participation in this study will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hepatic hemangioma, focal nodular hyperplasia, fatty liver, HBV infection, liver fibrosis, or cirrhosis who are undergoing hepatectomy or liver biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Change From Control in Liver Inflammation Degree at Postoperative | immediately after the surgery
  Postoperative liver tissue collection for the assessment of hepatic inflammation in participants.

SECONDARY OUTCOMES:
Change From Control in Hepatocyte Senescence Score at Postoperative | immediately after the surgery
  Postoperative liver tissue collection for the assessment of hepatocyte senescence in participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Nan, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No